CLINICAL TRIAL: NCT03404011
Title: Acute Effects of Propylene Glycol/Glycerol Intake on Cardiorespiratory Blood Parameters
Brief Title: Acute Effects of Propylene Glycol/Glycerol Intake on Blood Parameters
Acronym: AEPGGIBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Martin Chaumont, MD, Cardiology Fellow, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Université Libre de Bruxelles
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-10

CONDITIONS: Metabolic Complication
MeSH Terms: interventions — Propylene Glycol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propylene glycol and Glycerol intake (Experimental): One gram intake of a Propylene glycol/Glycerol mix (50:50)
  Interventions: Other: Propylene glycol and Glycerol intake
- Mimicking intake (Placebo Comparator): Mimicking Propylene glycol/Glycerol intake with the device turns off
  Interventions: Device: Mimicking intake

INTERVENTIONS:
Other: Propylene glycol and Glycerol intake — Intake of 1 gram of propylene glycol/Glycerol mix (50:50). Blood sample before, 5 minutes and 20 minutes after intake.
  Arms: Propylene glycol and Glycerol intake
Device: Mimicking intake — Mimicking propylene glycol/glycerol intake with the device turns off. Blood sample before, 5 minutes and 20 minutes after intake.
  Arms: Mimicking intake

SUMMARY:
The aim of this study is to evaluate the acute effect of propylene glycol and glycerol intake on cardiorespiratory blood parameters.

DETAILED DESCRIPTION:
Background : Propylene glycol/glycerol intake is increasingly popular. Acute effect of propylene glycol and glycerol intake on cardiorespiratory blood parameters is unknown. The investigators postulate that intake of propylene glycol and glycerol could modifiy cardiorespiratory blood parameters.

Aims of this study : to test the following hypotheses :

1) Acute intake of propylene glycol and glycerol modifies cardiorespiratory blood parameters.

To test this hypothesis, we will perform blood samples before and after intake of propylene glycol and glycerol. Participants will be tobacco smoker between 18 and 70 years old, with multiple cardiovascular risk factors, and who will undergo a cardiac catherization. After the cardiac catherization, the catheter will be used to perform serial blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Subject undergoing cardiac catherization
* Subject must be an active tobacco smoker

Exclusion Criteria:

* Symptoms of infection or inflammation
* Acute disease including heart rhythm disorder, acute coronary syndrome or decompensation of a chronic disease (heart failure, COPD,...)
* Unexpected and undesirable effects during the cardiac catherization procedure
* Respiratory failure requiring supplementary oxygen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory biological variables | 5 minutes
  Blood sample

SECONDARY OUTCOMES:
Cardiorespiratory biological variables | 20 minutes
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Martin Chaumont, MD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Saint-Pierre Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonnable request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03404011/Prot_SAP_001.pdf